CLINICAL TRIAL: NCT04191369
Title: A Randomized Controlled Trial Comparing Endoscopic Ultrasound Evaluation Versus Esophagogastroduodenoscopy in the Diagnosis of Portal Hypertension in Cirrhotic Patients
Brief Title: EGD vs EUS in Diagnosing Portal Hypertension in Cirrhotic Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EUS-EGD-PH
Record Dates: First submitted 2019-11-07; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Liver Cirrhoses; Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Endoscopy, Digestive System; Endosonography

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGD evaluation (Placebo Comparator): Esophogagastroduodenoscopy for the evaluation of esophageal varices, gastric varices and hypertensive gastropathy. Portal pressure gradient will be evaluated via interventional radiology as gold standard.
  Interventions: Diagnostic Test: Esophagogastroduodenoscopy
- EUS evaluation (Experimental): Endoscopic ultrasound evaluation for the presence of esophageal varices, peri and para-esophageal collateral veins, gastric varices, portal hypertensive gastropathy, azygos vein diameter, blood flow and BFVI.
  Portal pressure gradient will be evaluated via interventional radiology as gold standard.
  Interventions: Diagnostic Test: Endoscopic ultrasound

INTERVENTIONS:
Diagnostic Test: Esophagogastroduodenoscopy — Esophogagastroduodenoscopy for the evaluation of esophageal varices, gastric varices and hypertensive gastropathy. Portal pressure gradient will be evaluated via interventional radiology as gold standard.
  Arms: EGD evaluation
Diagnostic Test: Endoscopic ultrasound — Endoscopic ultrasound evaluation for the presence of esophageal varices, peri and para-esophageal collateral veins, gastric varices, portal hypertensive gastropathy, azygos vein diameter, blood flow and BFVI.
  Portal pressure gradient will be evaluated via interventional radiology as gold standard.
  Arms: EUS evaluation

SUMMARY:
Liver cirrhosis with the further development of portal hypertension implies structural and vasculature alteration in the portosplenic circulation.

Esophagogastroduodenoscopy is the standard of care for the detection and treatment of esophageal varices, as esophageal varices serve as a surrogate for estimating a portal pressure gradient > 10 mmHG.

Endoscopic ultrasound evaluation allows the detection of peri-esophageal collateral veins, perforating veins and para-esophageal collateral veins, which has demonstrated to be effective for the prediction of esophageal varices recurrence after variceal eradication.

The investigators aimed to compare esophagogastroduodenoscopy versus endoscopic ultrasound evaluation for the early diagnosis of portal hypertension in cirrhotic patients.

DETAILED DESCRIPTION:
A randomized control trial of 70 cirrhotic patients randomly submitted for esophagogastroduodenoscopy (35 patients) or EUS evaluation (35 patients) for the diagnosis of portal hypertension.

The portal pressure gradient will be defined based on portal vein catheterization via interventional radiology.

Esophagogastroduodenoscopy will evaluate the presence and grade of esophageal varices, presence and type of gastric varices, presence and signs of hypertensive gastropathy.

Endoscopic ultrasound will evaluate the presence of esophageal varices, the presence of gastric varices and the EUS- signs og hypertensive gastropathy, Azygos vein diameter, mean velocity and blood flow volume index.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Willingness to participate in the study
* Compensated liver cirrhosis based on clinical and imaging findings
* Written informed consent provided

Exclusion Criteria:

* Decompensated liver cirrhosis: ascitis, encephalopathy, gastrointestinal bleeding, infection
* Hemodynamic instability
* Pregant or nursing patients
* Patients with history of esophageal, gastric, liver, pancreas and spleen tumors
* Severe uncontrolled coagulopathy
* Any contraindication for portal pressure gradient meassurement via radiological evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of portal hypertension | During portal pressure gradient meassurement up to 4 weeks after randomization
  Portal hypertension diagnosis based on portal pressure gradient

SECONDARY OUTCOMES:
diagnostic accuracy of esophagogastroduodenoscopy | during esophagogastroduodenoscopy procedure up to 2 weeks after randomization
  Overall accuracy of esophagogastroduodenoscopy in the detection and grading of esophageal varices, gastric varices and hypertensive gastropathy.
diagnostic accuracy of endoscopic ultrasound | during endoscopic ultrasound evaluation up yo 2 weeks after randomization
  Overall accuracy of endoscopc ultrasound evaluation in the detection and grading of esophageal varices, gastric varices and hypertensive gastropathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boustiere C, Dumas O, Jouffre C, Letard JC, Patouillard B, Etaix JP, Barthelemy C, Audigier JC. Endoscopic ultrasonography classification of gastric varices in patients with cirrhosis. Comparison with endoscopic findings. J Hepatol. 1993 Sep;19(2):268-72. doi: 10.1016/s0168-8278(05)80581-1. PMID 8301060
- [Background] Hammoud GM, Ibdah JA. Utility of endoscopic ultrasound in patients with portal hypertension. World J Gastroenterol. 2014 Oct 21;20(39):14230-6. doi: 10.3748/wjg.v20.i39.14230. PMID 25339809